CLINICAL TRIAL: NCT03246763
Title: Active Recreation Through Community-Healthcare Engagement Study
Acronym: ARCHES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00084070
Record Dates: First submitted 2017-08-04; First posted 2017-08-11 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Childhood Obesity; Quality of Life
Keywords: childhood obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a mixed-methods study using focus groups and interviews to explore the facilitators and barriers to program implementation, and a time-series analysis to examine program engagement and individual health outcomes. This study design will be repeated at each of the four sites. Aim 1 will consent and enroll program providers to obtain qualitative feedback on program design and implementation; Aim 2 will collect de-identified program-level data on attendance and program components; Aim 3 will consent patients for individual-level baseline and outcomes data.Subjects will be enrolled at our community sites. A research assistant will conduct all the enrollment, consent, and data collection. Where needed, the investigators will report or obtain required IRB authorization agreements for each site, including Federal Wide Assurances, Data Transfer Agreements, or other documents as required by federal regulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Durham County (Experimental): The intervention will include nutrition and fitness programming at a community center. The program will be open at least two sessions per week, each session lasting at least 1 hour. The program coordinator will run the programming, which will consist of comprehensive wellness activities. Each session will include at least 60 minutes of exercise and/or active play, and each session will have an additional special "theme." For example, one session might include a cardio focused class, and one session might include a yoga class. The number and which sessions the participants attend each week is voluntary; clinic staff will recommend participation in as many sessions per week as possible. Participation is voluntary, and patients may opt-out at any time. Participants will be told that they can indicate to their provider or the program coordinator at any time either by phone or during the clinic appointment that they wish to opt-out of the study and its assessments.
  Interventions: Behavioral: Integrated community-healthcare childhood obesity treatment
- Richmond/Montgomery Counties (Experimental): The intervention will include nutrition and fitness programming at a community center. The program will be open at least two sessions per week, each session lasting at least 1 hour. The program coordinator will run the programming, which will consist of comprehensive wellness activities. Each session will include at least 60 minutes of exercise and/or active play, and each session will have an additional special "theme." For example, one session might include a cardio focused class, and one session might include a yoga class. The number and which sessions the participants attend each week is voluntary; clinic staff will recommend participation in as many sessions per week as possible. Participation is voluntary, and patients may opt-out at any time. Participants will be told that they can indicate to their provider or the program coordinator at any time either by phone or during the clinic appointment that they wish to opt-out of the study and its assessments.
  Interventions: Behavioral: Integrated community-healthcare childhood obesity treatment
- TBD (Experimental): The intervention will include nutrition and fitness programming at a community center. The program will be open at least two sessions per week, each session lasting at least 1 hour. The program coordinator will run the programming, which will consist of comprehensive wellness activities. Each session will include at least 60 minutes of exercise and/or active play, and each session will have an additional special "theme." For example, one session might include a cardio focused class, and one session might include a yoga class. The number and which sessions the participants attend each week is voluntary; clinic staff will recommend participation in as many sessions per week as possible. Participation is voluntary, and patients may opt-out at any time. Participants will be told that they can indicate to their provider or the program coordinator at any time either by phone or during the clinic appointment that they wish to opt-out of the study and its assessments.
  Interventions: Behavioral: Integrated community-healthcare childhood obesity treatment
- To be determined (Experimental): The intervention will include nutrition and fitness programming at a community center. The program will be open at least two sessions per week, each session lasting at least 1 hour. The program coordinator will run the programming, which will consist of comprehensive wellness activities. Each session will include at least 60 minutes of exercise and/or active play, and each session will have an additional special "theme." For example, one session might include a cardio focused class, and one session might include a yoga class. The number and which sessions the participants attend each week is voluntary; clinic staff will recommend participation in as many sessions per week as possible. Participation is voluntary, and patients may opt-out at any time. Participants will be told that they can indicate to their provider or the program coordinator at any time either by phone or during the clinic appointment that they wish to opt-out of the study and its assessments.
  Interventions: Behavioral: Integrated community-healthcare childhood obesity treatment

INTERVENTIONS:
Behavioral: Integrated community-healthcare childhood obesity treatment — The intervention will include nutrition and fitness programming at a local community center. The program will be open at least two sessions per week, each session lasting at least 1 hour. The program coordinator will run the programming, which will consist of wellness activities. Each session will include at least 60 minutes of exercise and/or active play, and each session will have an additional special "theme." For example, one session might include a cardio focused class, and one session might include a yoga class. The number and which sessions the participants attend each week is voluntary; clinic staff will recommend participation in as many sessions per week as possible. Participation is voluntary, and patients may opt-out at any time. Participants will be told that they can indicate to their provider or the program coordinator at any time either by phone or during the clinic appointment that they wish to opt-out of the study and its assessments.

SUMMARY:
Current obesity treatment guidelines recommend 26 or more hours of behavior treatment, delivered over a 6-month period in a multidisciplinary weight management clinic. However, this guideline is not feasible in real-world clinic settings where medical visits are costly and poorly reimbursed, and attrition is high, particularly among the most vulnerable children. The National Collaborative on Child Obesity Research has issued a call for research investigating healthcare-community partnerships to improve the effectiveness of child obesity treatment. The World Health Organization supports this approach, and in 2015 modified the chronic disease model to include healthcare-community integration. ARCHES is a three-year project that will develop and evaluate an effective, engaging, and scalable community-healthcare treatment option for low-income and racially diverse children. The project engages four communities in North Carolina and facilitates a local clinic-community partnership, supports the development of an integrated childhood obesity treatment program, and evaluates the feasibility of the integrated program model. The effectiveness of the integrated model will also be evaluated, as we will monitor patient outcomes associated with participation. Participation among teens (ages 11-18) will be incentivized where teen/caregiver dyads will be randomized to a gain or loss frame group at the beginning of the study and have the opportunity to receive and redeem points for attending sessions. Patient and process outcomes associated with participation in the integrated model with and without financial incentives will be evaluated.

DETAILED DESCRIPTION:
The investigators propose a three-year project to evaluate the implementation feasibility and effectiveness of an integrated clinic-community model of child obesity treatment. The investigators will engage four communities in North Carolina, facilitate a local clinic-community partnership, support the development of an integrated child obesity treatment program, and monitor outcomes. To evaluate implementation feasibility the investigators will measure fidelity, reach, acceptability, uptake and cost. To evaluate the program model the investigators will conduct a classical program evaluation by monitoring aggregate referral, enrollment and attendance data, as well as safety and patient satisfaction. To report patient outcomes associated with participation in the integrated model, the investigators will measure participant-level outcomes over a 6-month period, including changes in nutrition and physical activity behaviors, quality of life, cardiovascular fitness, and body mass index.

ELIGIBILITY:
Sampling:

- Patients enrolled by their physician in the clinic-community program

Inclusion:

* Child aged 2-17 years
* Child with age- and gender-specific BMI ≥ 85th percentile

Exclusion:

* Inability to read and write in English or Spanish
* Parent with severe medical or mental health condition limiting ability to attend appointments
* Child with severe medical or mental health condition limiting ability to attend appointments or participate in behavioral therapies
* Parent and child live greater than 50 miles from the clinic and community center
* Plan to move out of state in the next 6 months, or plan to live in another state for 2 months or longer within the next 6 months (ex., summer vacation).
* Child with medical condition as cause of obesity (e.g., hypothyroidism, Cushing's Syndrome, Prader-Willi Syndrome, drug-induced obesity)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 202 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Eligibility | Baseline
  Number of eligible patients
Referral | Baseline
  Number of referred patients
Enrollment | Baseline
  Number of patients referred who enroll
Attendance | Through study completion, average of 1 year
  Number of participants present at each activity session
Fidelity | Through study completion, average of 1 year
  Measured by program post-session evaluation survey
Change in quality of life | Baseline, 6 months, 12 months
  Measured by Sizing me Up survey
Change in height | 0 months, 3 months, 6 months, 12 months
Change in nutrition habits (self report) | 0 months, 3 months, 6 months, 12 months
Food insecurity | Baseline
  Measured by The Hunger Vital Sign food insecurity assessment
Change in cardiovascular fitness | 0 months, 3 months, 6 months
Patient satisfaction | 6 months
  Measured by patient satisfaction survey
Change in social cohesion | 3 months, 6 months
  Measured by social cohesion questionnaire
Change in weight | 0 months, 3 months, 6 months, 12 months
Change in activity (self report) | 0 months, 3 months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - First Health, Biscoe, North Carolina
  - East Durham Children's Initiative, Durham, North Carolina
  - Duke Healthy Lifestyles, Durham, North Carolina
  - Better Health, Fayetteville, North Carolina
  - Goldsboro Parks and Recreation, Goldsboro, North Carolina
  - Wake Med, Raleigh, North Carolina
  - Healthy Rowan, Salisbury, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alexander E, Skinner A, Gaskin K, Jones J, Wong C, Loflin C, Fleming R, Howard J, Armstrong S, Neshteruk C. A Mixed-Methods Examination of Referral Processes to Clinic-Community Partnership Programs for the Treatment of Childhood Obesity. Child Obes. 2021 Dec;17(8):516-524. doi: 10.1089/chi.2020.0361. Epub 2021 Jul 5. PMID 34227849